CLINICAL TRIAL: NCT02718820
Title: Immunomodulation of Pembrolizumab Plus Docetaxel for the Treatment of Recurrent or Metastatic (R/M) Squamous Cell Carcinoma of the Head and Neck (HNSCC) After Platinum Failure
Brief Title: Pembrolizumab Plus Docetaxel for the Treatment of Recurrent or Metastatic Head and Neck Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Thorsten Fuereder, Assoc.Prof.PD.Dr., Medical University of Vienna
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PemDoc II
Record Dates: First submitted 2016-03-15; First posted 2016-03-24 (Estimated); Results first posted 2023-12-04 (Actual); Last update posted 2024-01-09 (Actual); Status verified 2023-12

CONDITIONS: Head and Neck Carcinoma
MeSH Terms: interventions — Docetaxel; pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Docetaxel plus pembrolizumab (Experimental): Docetaxel 75mg/m2 plus pembrolizumab 200mg will be administered every 3 weeks intravenously for 6 cycles. Thereafter pembrolizumab 200mg every 3 weeks will be given as maintenance therapy until progression.
  Interventions: Drug: Docetaxel; Drug: Pembrolizumab

INTERVENTIONS:
Drug: Docetaxel — Docetaxel 75mg/m2; q21
  Other Names: Taxotere
Drug: Pembrolizumab — Pembrolizumab 200mg, q21
  Other Names: Keytruda

SUMMARY:
Squamous cell carcinoma of the head and neck, which accounts for 90% of head and neck cancers, is the tenth most common cancer worldwide with over 650000 new cases per year. The major risk factors for HNSCC development comprise alcohol and tobacco consumption. During the last decades human papilloma virus infection (HPV) has been identified to contribute to the development of oropharyngeal HNSCC in a subgroup of patients5. Standard treatment options include surgery, (chemo)radiation and chemotherapy. Despite improvements of treatment regimens the recurrence rate of stage III/IV disease after curative therapy is about 30-40%. In locoregionally unresectable recurrent or metastatic disease palliative poly-chemotherapy is the mainstay of therapy.The median survival time of these patients is 6-8 months. Based on the results of the EXTREME study a combination regimen containing a platinum drug, 5 fluorouracil (5-FU) and weekly cetuximab has become standard of care in this setting. For patients, who progressed after platinum based therapy, treatment options are scarce. Besides platinum drugs, taxanes such as paclitaxel or docetaxel were shown to be of particular use in this setting. Apart from that there has been increasing preclinical and clinical evidence that immune-checkpoint inhibitors such as pembrolizumab might play a role in HNSCC. Thus, it is the aim of this study to test if the combination of docetaxel and pembrolizumab after platinum failure is an effective and safe regimen.

DETAILED DESCRIPTION:
not provided

ELIGIBILITY:
Inclusion Criteria:

* The patient has provided written informed consent prior to any study-related procedure.
* The patient is at least 18 years of age
* Histologically proven locally advanced unresectable, recurrent and/or metastatic squamous cell carcinoma of the oropharynx, hypopharynx, larynx or oral cavity not amenable for salvage surgery
* P16 mutation status has to be determined
* Documented progressive disease based on investigator assessment according to RECIST 1.1, following receipt of a cisplatin and/or carboplatin based regimen independent of whether patient progressed during or after platinum based therapy. Platinum therapy might have been administered either as part of induction chemotherapy (12 months), chemoradiation (6 months) or as first line systemic palliative chemotherapy (6 months).
* Measurable disease according to RECIST 1.1.
* The patient has a life expectancy of at least 3 months.
* Has a performance status of 0 or 1 on the Eastern Cooperative Oncology Group (ECOG) Performance Scale
* Female subject of childbearing potential should have a negative urine or serum pregnancy prior to study registration and re-tested within 72 hours prior to receiving the first dose of study medication. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
* Female subjects of childbearing potential should be willing to use 2 methods of birth control or be surgically sterile, or abstain from heterosexual activity for the course of the study through 120 days after the last dose of study medication. Subjects of childbearing potential are those who have not been surgically sterilized or have not been free from menses for > 1 year.
* Male subjects should agree to use an adequate method of contraception starting with the first dose of study therapy through 120 days after the last dose of study therapy.
* Demonstrate adequate organ function as defined in Table 1, all screening labs should be performed within 10 days of treatment initiation.

Exclusion Criteria:

* Prior taxane therapy is not allowed except as part of induction therapy (at least 6 months before study entry)
* Nasopharyngeal carcinomas or salivary glands cancers are not eligible
* Is currently participating and receiving study therapy or has participated in a study of an investigational agent and received study therapy or used an investigational device within 4 weeks of the first dose of treatment.
* Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of trial treatment.
* Has a known history of active Bacillus Tuberculosis (TB)
* Hypersensitivity to pembrolizumab or any of its excipients.
* Has had a prior anti-cancer monoclonal antibody (mAb) within 4 weeks prior to study Day 1 or who has not recovered (i.e., ≤ Grade 1 or at baseline) from adverse events due to agents administered more than 4 weeks earlier.
* Has had prior chemotherapy, targeted small molecule therapy, or radiation therapy within 2 weeks prior to study Day 1 or who has not recovered (i.e., ≤ Grade 1 or at baseline) from adverse events due to a previously administered agent.
* Note: If subject received major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting therapy.
* Has a known additional malignancy that is progressing or requires active treatment. Exceptions include basal cell carcinoma of the skin or squamous cell carcinoma of the skin that has undergone potentially curative therapy or in situ cervical cancer.
* Has known active central nervous system (CNS) metastases and/or carcinomatous meningitis. Subjects with previously treated brain metastases may participate provided they are stable (without evidence of progression by imaging for at least four weeks prior to the first dose of trial treatment and any neurologic symptoms have returned to baseline), have no evidence of new or enlarging brain metastases, and are not using steroids for at least 7 days prior to trial treatment. This exception does not include carcinomatous meningitis which is excluded regardless of clinical stability.
* Has active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (e.g. thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.
* Has known history of, or any evidence of active, non-infectious pneumonitis.
* Has an active infection requiring systemic therapy.
* Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
* Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
* Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the pre-screening or screening visit through 120 days after the last dose of trial treatment.
* Has received prior therapy with an anti-PD-1, anti-PD-L1, or anti-PD-L2 agent.
* Has a known history of Human Immunodeficiency Virus (HIV) (HIV 1/2 antibodies).
* Has known active Hepatitis B (e.g., HBsAg reactive) or Hepatitis C Virus (HCV) RNA [qualitative] is detected.
* Has received a live vaccine within 30 days of planned start of study therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2016-03; Primary Completion 2021-12 (Actual); Study Completion 2021-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thorsten Fuereder, MD, Principal Investigator — Medical University of Vienna
Locations (1):
- Medical University of Vienna, Vienna, Austria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Fullt text of the published manuscript — https://doi.org/10.1016/j.oraloncology.2021.105634

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Docetaxel Plus Pembrolizumab
Started | 22
Completed | 22
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: 22
Arm/Group | Docetaxel Plus Pembrolizumab
Number analyzed (Participants) | 22
Age, Customized [Median (Full Range); unit: years] | 62.5 [44 to 78]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 18
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 22
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  Austria | 22

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate
Description: Overall response rate will be measured
Time Frame: 1 year
Measure: Mean (95% Confidence Interval); unit: percentage
Arm/Group | Docetaxel Plus Pembrolizumab
Number analyzed (Participants) | 22
percentage | 22.7 [10.1 to 43.3]

2. Secondary Outcome: Median Overall Survival (OS)
Description: Kaplan meier curves will be calculated and OS in months measured
Time Frame: 4 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Docetaxel Plus Pembrolizumab
Number analyzed (Participants) | 22
months | 21.3 [6.3 to 31.3]

3. Secondary Outcome: Treatment-related Adverse Events
Description: Number of participants with treatment-related adverse events as assessed by CTCAE v4.0
Time Frame: 4 years
Measure: Number; unit: Count of Participants
Arm/Group | Docetaxel Plus Pembrolizumab
Number analyzed (Participants) | 22
Count of Participants | 22

4. Secondary Outcome: Median Progression Free Survival (PFS)
Description: Kaplan meier curves will be calculated and PFS in months measured
Time Frame: 4 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Docetaxel Plus Pembrolizumab
Number analyzed (Participants) | 22
months | 5.8 [2.7 to 11.6]

ADVERSE EVENTS:
Time Frame: 5 years
Arm/Group | Docetaxel Plus Pembrolizumab
All-Cause Mortality (participants affected / at risk) | 17/22
Serious Adverse Events (participants affected / at risk) | 12/22
Other Adverse Events (participants affected / at risk) | 22/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Docetaxel Plus Pembrolizumab (N=22)
Thrombocytopenia (Blood and lymphatic system disorders) | 1
Febrile Neutropenia (Blood and lymphatic system disorders) | 1
Decreased General Condition (General disorders) | 4
Nausea (Gastrointestinal disorders) | 1
Oral hemorrhage (Gastrointestinal disorders) | 5
Lung Infection (Infections and infestations) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Docetaxel Plus Pembrolizumab (N=22)
Febrile Neutropenia (Blood and lymphatic system disorders) | 3
Anemia (Blood and lymphatic system disorders) | 9
Neutropenia (Blood and lymphatic system disorders) | 15
Nausea (Gastrointestinal disorders) | 3
Dysphagia (Gastrointestinal disorders) | 1
Oral hemorrhage (Gastrointestinal disorders) | 3
Gastric hemorrhage (Gastrointestinal disorders) | 3
Dehydration (Metabolism and nutrition disorders) | 2
Hypophosphatemia (Metabolism and nutrition disorders) | 1
Creatinine increased (Investigations) | 1
GGT increased (Investigations) | 2
Syncope (Nervous system disorders) | 2
Lung infection (Infections and infestations) | 1
Sepsis (Infections and infestations) | 1
Wound infection (Infections and infestations) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-06-15): https://cdn.clinicaltrials.gov/large-docs/20/NCT02718820/Prot_SAP_000.pdf